CLINICAL TRIAL: NCT03343912
Title: Dose-response Study With Three Vaginal Rings With Different Doses of Estriol and Trimegestone: Effect on Progesterone and Estradiol Levels in Healthy Females With Childbearing Potential
Brief Title: Estriol and Trimegestone Dose-response Trial With Single Dose Application of Vaginal Rings
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galeno Desenvolvimento de Pesquisas Clínicas (Other Government)
Collaborators: SocraTec R&D GmbH (Other)
Responsible Party: Principal Investigator, Gilberto De Nucci, Director, Galeno Desenvolvimento de Pesquisas Clínicas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GDN 012/17
Record Dates: First submitted 2017-11-07; First posted 2017-11-17 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Pregnancy
Keywords: Estriol; Trimegestone; Vaginal Ring
MeSH Terms: interventions — Estriol; trimegestone

STUDY DESIGN:
Intervention Model Description: Single centre, open-label, randomized (assignment to treatment group), parallel-group, three-arm single-dose clinical trial with application performed over 1 treatment cycle of 21 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test 1 vaginal ring (Experimental): Single intravaginal application of 1 vaginal ring of Estriol 0.400 mg/day and Trimegestone 0.06 mg/day (Test 1) over 21 days
  Interventions: Drug: Estriol 0.400 mg/day and Trimegestone 0.06 mg/day
- Test 2 vaginal ring (Experimental): Single intravaginal application of 1 vaginal ring of Estriol 0.300 mg/day and Trimegestone 0.12 mg/day (Test 2) over 21 days
  Interventions: Drug: Estriol 0.300 mg/day and Trimegestone 0.12 mg/day
- Test 3 vaginal ring (Experimental): Single intravaginal application of 1 vaginal ring of Estriol 0.200 mg/day and Trimegestone 0.18 mg/day (Test 3) over 21 days
  Interventions: Drug: Estriol 0.200 mg/day and Trimegestone 0.18 mg/day

INTERVENTIONS:
Drug: Estriol 0.400 mg/day and Trimegestone 0.06 mg/day — Vaginal ring with a nominal delivery rate of 0.400 mg/d estriol (E3) and 0.06 mg/d trimegestone (TMG), vaginal application
  Arms: Test 1 vaginal ring
Drug: Estriol 0.300 mg/day and Trimegestone 0.12 mg/day — Vaginal ring with a nominal delivery rate of 0.300 mg/d estriol (E3) and 0.12 mg/d trimegestone (TMG), vaginal application
  Arms: Test 2 vaginal ring
Drug: Estriol 0.200 mg/day and Trimegestone 0.18 mg/day — Vaginal ring with a nominal delivery rate of 0.200 mg/d estriol (E3) and 0.18 mg/d trimegestone (TMG), vaginal application
  Arms: Test 3 vaginal ring

SUMMARY:
This clinical trial is performed as proof of pharmacological action investigation by demonstration of ovulation inhibition (dose-response study) under treatment with three Test vaginal rings releasing varying doses of estriol (E3) and trimegestone (TMG).

Blood samples for determination of estradiol (E2) and progesterone (PG) levels will serve as pharmacodynamic surrogate parameters for characterization of the treatment effect on the endogenous hormones.

Blood samples for determination of E3 and TMG in plasma will be collected in order to characterize pharmacokinetic parameters.

Additionally, local tolerability characterized by gynecological inspection of the vaginal mucosa prior to and after insertion of the Investigational Medicinal Product (IMPs) is planned to be assessed

DETAILED DESCRIPTION:
The IMPs, releasing either 0.400 mg E3 and 0.06 mg TMG, or 0.300 mg E3 and 0.12 mg TMG, or 0.200 mg E3 and 0.18 mg TMG per 24 h, will be applied intravaginally and remain in the vagina for the subsequent 21 days (single dose, 1 treatment cycle). A total of 36 female subjects, 12 per treatment group, are intended to be randomized.

Blood samples for determination of E2 and PG levels will be collected during treatment and until 20 days after removal of the ring. Blood samples for determination of E3 and TMG in plasma will be collected over the treatment period and until 48 h after removal of the ring.

Bleeding intensity will also be documented during treatment and until 20 days after removal of the vaginal ring in a diary to characterize the effects of the different treatments.

ELIGIBILITY:
Inclusion Criteria:

* Under treatment with a commercially available combined oral contraceptive containing 30 µg ethinylestradiol (EE) and 150 µg levonorgestrel (LVN) for the last 3 months prior to enrolment
* Body-mass index (BMI): ≥ 18.5 kg/m² and ≤ 30.0 kg/m²
* Good state of health
* Non-smoker, ex-smoker for at least 3 months
* Regular menstrual cycle with a length between 21 and 35 days
* Written informed consent, after having been informed about benefits and potential risks of the clinical trial

Exclusion Criteria:

* Existing diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the IMPs
* Subjects with severe allergies or multiple drug allergies
* Positive anti human immunodeficiency virus (anti-HIV) test, hepatitis B surface antigen (HBs-AG) test or anti hepatitis C virus (anti-HCV) test
* Presence or history of venous or arterial thrombosis, cerebrovascular accident, or increased risk of thrombosis
* Diabetes mellitus
* Unclarified vaginal bleeding or frequent infections of the urogenital tract
* Severe or chronic constipation
* Presence or history of migraine
* Drug or alcohol dependence
* Blood donation or other blood loss of more than 400 ml within the last 3 months
* Participation in a clinical trial during the last 6 months
* Pregnant or lactating women
* Subjects who do not agree to apply a barrier method for contraception

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Measurement of E2 and PG plasma levels | 0 - 41 days
  Blood sampling for the determination of plasma levels of E2 and PG, in participants of each treatment group, as surrogate variables for treatment response.
Measurement of E3 and TMG plasma levels | 0 - 23 days
  Blood sampling for the determination of plasma levels of E3 and TMG, in participants of each treatment group.

SECONDARY OUTCOMES:
Bleeding intensity | start of treatment until 42 days after treatment
  Bleeding intensity, graded as "no bleeding", "spotting" or "bleeding" as recorded in diary by the subject on a daily basis
Number of adverse events per participant | up to 42 days after treatment
  Number of adverse events, in each treatment group, including clinically relevant alterations of vital signs and laboratory tests results
Maximum Plasma Concentration (Cmax) of E3 and TMG | 0 - 23 days
  Determination of Cmax for E3 and for TMG, based on plasma concentrations of samples obtained.
Area Under the Curve (AUC) for E3 and TMG | 0 - 23 days
  Calculation of the AUC for E3 and for TMG, based on plasma concentrations of samples obtained

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto De Nucci, MD, Principal Investigator — Galeno Desenvolvimento de Pesquisas Clinicas Ltda. - ME
Locations (1):
- Galeno Desenvolvimento de Pesquisas Clinicas Ltda. - ME, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No